CLINICAL TRIAL: NCT05271851
Title: PEP (Parent and Child-Informed, Environmentally-Responsive Pediatric Asthma) Study
Brief Title: Tailoring Mindfulness Interventions for Families Managing Chronic Health Conditions
Acronym: PEP
Status: Completed | Type: Observational
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Wisconsin, Madison (Other); University of Maryland, Baltimore (Other); University of Memphis (Other)
Responsible Party: Sponsor
Other Study IDs: AT010207
Record Dates: First submitted 2022-02-27; First posted 2022-03-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Mindfulness; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is not an intervention or treatment study. It is an observational qualitative data study about tailoring a mindfulness intervention to assist families managing chronic health conditions.

DETAILED DESCRIPTION:
This is not an intervention or treatment study. It is an observational qualitative data study. Collecting information from virtual audio only interviews from between 30 and 40 US adults about whether a mindfulness intervention would assist families managing chronic health conditions; and if so, how should it be tailored to meet their needs.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and either a long-time mindfulness practitioner/instructor or an adult managing a chronic health condition for yourself or a close family member

Exclusion Criteria:

* unable to complete an audio interview in English lasting 30-60 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: English speaking and either a long-time mindfulness practitioner/instructor or an adult managing a chronic health condition for yourself or a close family member
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
what families managing chronic illness want in a mindfulness intervention | 30 to 60 minute interview
  structured open ended questions analyzed with grounded theory- no quantitative data will be captured

CONTACTS AND LOCATIONS:
Overall Officials: Robin Puett, PhD, Principal Investigator — UMD
Locations (1):
- UMD, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No